CLINICAL TRIAL: NCT02405559
Title: The Occlusion Pressure of Superficial Lymphatics in the Lower Extremity of Healthy Volunteers: A Near Infrared Lymphofluoroscopy Approach
Brief Title: Lymphatic Occlusion Pressure in Lower Limb
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Centre Hospitalier Universitaire Saint Pierre (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: Ly-Occl-Pressure-2
Record Dates: First submitted 2015-03-05; First posted 2015-04-01 (Estimated); Last update posted 2015-04-01 (Estimated); Status verified 2015-03

CONDITIONS: Lymphatic Function
MeSH Terms: interventions — Indocyanine Green

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Lymphatic occlusion pressure lower limb (Experimental): injection of 100µg Indocyanine Green in the first interdigital space and application of increasing pressure around the leg to visualize at which pressure lymph flow is interrupted.
  Interventions: Drug: Indocyanine Green

INTERVENTIONS:
Drug: Indocyanine Green — Intradermal injection of Indocyanine Green in the first interdigital space of the studied leg
  Other Names: ICG

SUMMARY:
The lymphatic system is one of the keystones of fluid homeostasis in the interstitium. In analogy with the arterial systolic pressure, the lymphatic pressure can give us information about the functioning of the cardiovascular system and fluid exchange. Actually, knowledge about this physiological parameter is incomplete because of the lack of technology. Former measurement techniques of the lymphatic pressure in the living healthy man were invasive and too complex to be interpreted.

The lymphatic occlusion pressure has to be clarified because lymphedema treatment, concerning the pressure to be applied on the edematous tissue is still based on controversial concepts.

On one hand, techniques such as Manual Lymphatic Drainage, sustain the necessity to apply a very low pressure in order to avoid the squeezing of superficial lymph vessels. On the other hand sustainers of Intermittent Compression Therapy advocate the necessity to apply relatively high pressure to obtain a decongesting effect. These completely opposite opinions triggered us to study lymphatic pressure more thoroughly.

Lymphofluoroscopy (emerging imaging technique in the field of lymphology) is now used since 3 years by the promoters of this study to visualize the architecture of the superficial lymphatic network and the progression of the lymph inside the highlighted vessels. This technique will be used in the present (prospective and multicentric) study to observe the effect of a pressure applied on the lower limb on the displacement of the lymph, and then to determine the occlusion pressure of the lymphatic vessels. The investigators already studied the occlusion pressure of the superficial lymphatic vessels of the upper limb in a previous study. The investigators would like to complete our results with the lower limb.

DETAILED DESCRIPTION:
Injection of contrast agent:

Indocyanine Green (ICG) is a tricarbocyanine dye that is commonly used for hepatic, cardiovascular, plastic surgery and ophthalmology applications. It is usually injected intravenously at a dose comprised between 0.1 and 0.5 mg/kg. After administration, ICG binds to plasmatic proteins, lipoproteins and lipids, and is thereafter rapidly and completely cleared from blood by the liver. ICG is excited and emits fluorescence in the near-infrared (around 800 nm).

In this study, the investigators will suspend ICG in 25 ml pure water and subsequently diluted with pure water to reach a final concentration of 0.2 mg/ml. Each subject will receive an intradermal injection of 0.5 ml of diluted ICG (e.i. 100µg), using a hypodermic needle. The investigators will standardize the injection point and inject ICG intradermally in the first interdigital space, according to the injection method used for lymphoscintigraphy. In this way, the investigators highlight systematically the same area of the superficial lymphatic network.

Fluorescence images acquisition:

After injection, the injection sites will be covered with tape to avoid camera oversaturation, and to avoid spreading of ICG on the skin and undesirable fluorescent background on the images. To obtain fluorescence imaging of leg lymphatic flow, a near-infrared fluorescence imaging system will be used (Photo Dynamic Eye, or PDE camera from Hamamatsu Photonics - Japan). The camera is maintained in a fix position, 15 cm above the investigation field, by a holding system from Noga Tools. The amplified analogic signal is transformed into a digital signal by a converter from Terratec (Model Grabster AV 450 MX) and transferred to a monitor, which allows to visualize lymphatic network and lymph flow in real-time. Images will be recorded on a dedicated external hard disk drive Iomega, model MDHDU.

The session will take place in a dark room, to allow NIR fluorescence images acquisition.

Specific manual lymphatic drainage, developed by the first author and his team under NIRF feedback, is performed immediately after the injection, during the whole experimental session in order to be sure that the examined lymphatic vessels permanently contain lymph. The lymph is propelled with the hand of the operator from the injection point to a limit line drawn on the skin at 5 cm before the distal extremity of the transparent cuff. This optimized manual lymphatic drainage will be performed for 3 minutes in order to easily detect the superficial lymphatic vessels at the distal region of the leg and to mark the area of interest. The MLD is standardized by the first author for this experiment, and composed by a continuous and repeated sequence, executed from distal to proximal, of 3 "fill up" maneuvers realized on the injection point, succeeded by 2 "wash out" maneuvers realized from the injection point to the limit line before the cuff. Then, two fluorescent lines are drawn on the skin in a distance of 50 mm in order to limit the space of reference.

The cuff of the transparent sphygmomanometer is placed on the distal part of the leg, just above the ankle.

The sphygmomanometer is connected to a pressure meter, indicating mm of Mercury (Testo® 510 Digital Manometer precision 0.1mmHg.).

The PDE camera will be maintained perpendicularly on the major axis of the leg, at the level of the middle of the cuff.

In order to make sure that observed lymphatic vessels contain lymph, the fluorescent lymph is propelled during all the experience with the hand of the operator from the injection point to a limit line drawn on the skin at 5 cm before the distal extremity of the transparent cuff.

* First step: as baseline we record and observe the lymphatic flow under the un-inflated cuff.
* Second step: the cuff is inflated at 30mmHg, images are recorded during three lymph flow passages.

Three independent observers are present. They control the three passages of lymph in order to give the consent to go over to the next pressure step.

- Third step: The investigators increase the inflated pressure in steps of 10 mmHg recording images at each increase (waiting for three passages of lymph at each step).

The experiment is completed as soon as the investigators visually note the complete stop of lymph progression under the transparent cuff. At that moment, the pressure is reduced by 10mmHg in order to validate the return of the lymph flow. After this step, the investigators observe and record images of the lymphatic vessel from the injection point up to the root of the limb.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers
* Written informed consent signed

Exclusion Criteria:

* Coronary disease
* Pregnancy
* Allergy to iodine or to shellfish
* Breastfeeding
* Advanced renal impairment
* Minors
* Thyroid pathology
* Primary and secondary lymphedema anywhere on the body
* Oncologic history
* Familial lymphedema
* Previous surgery on the studied member, causing risk of a subclinical lymphedema

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2015-05; Primary Completion 2015-12 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Lymph flow active or not, depending on the pressure applied | 1 minute
  The sphygmomanometer is connected to a pressure meter, indicating mm of Mercury (Testo® 510 Digital Manometer precision 0.1mmHg.).

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Paul Belgrado, Principal Investigator — CHU St-Pierre
Locations (1):
- CHU St-Pierre - Lymphology Clinic of Brussels, Brussels, Belgium